CLINICAL TRIAL: NCT00640562
Title: Comparison of Quetiapine Extended-Release (Seroquel XR™) and Risperidone in the Treatment of Depressive Symptoms, in Schizophrenic or Schizoaffective Patients: A Randomized, Open Label, Flexible-dose, Parallel Group, Non Inferiority, 12-week Study
Brief Title: Quetiapine Extended Release Depression Symptoms
Acronym: ExAttitude
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00031
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Results first posted 2012-06-19 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-05

CONDITIONS: Schizophrenia; Depression
Keywords: Schizophrenia; Depression; Quetiapine
MeSH Terms: conditions — Schizophrenia; Depression | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quetiapine Extended Release (Experimental)
  Interventions: Drug: Quetiapine Extended Release
- Risperidone (Active Comparator)
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Quetiapine Extended Release — Uptitrated starting from 300 mg in the evening on day 0, then increasing to 600 mg and up to 800 mg in the following two evenings. Previous antipsychotic was taken at the full dose on day 0, half dose on day 1 and stopped from day 2. From day 3 onwards it was possible to adjust the Seroquel XR dose, depending on the clinical response and tolerability of the patient, within the range of 400-800 mg per day
  Other Names: Seroquel XR™
  Arms: Quetiapine Extended Release
Drug: Risperidone — Uptitrated starting from 1 mg bid (morning and evening) on day 0, then increasing to 2 mg bid and up to 3 mg in the following two days. As per the other arm, previous antipsychotic was taken at the full dose on day 0, half dose on day 1 and stopped from day 2. From day 2 onwards, it was allowed to adjust he dose of Risperidone depending on the clinical response and tolerability of the patient.
  Other Names: Risperdal
  Arms: Risperidone

SUMMARY:
Aim of the study is to assess if the new compound Seroquel XR™ is non-inferior to Risperidone, considered as the reference drug for the treatment of depressive symptoms of schizophrenia.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Patients who satisfy the criteria for diagnosis of schizophrenia or schizoaffective disorder according to DSM-IVTR
* Baseline depressive symptoms, assessed by means of HAM-D (21-item) score ≥20, and HAM-D item 1 score ≥2

Exclusion Criteria:

* Any DSM-IV Axis I disorder other than schizophrenia and schizoaffective disorder
* Patients treated with depot antipsychotic medications within 1 dosing interval before day 0; patients treated with other AP oral medications during the trial except for the switch period
* Use of Clozapine within 28 days prior to enrollment or Clozapine non responders
* Any significant clinical disorder that, in the opinion of the investigator, made the subject unsuitable to be given treatment with an investigational drug
* An absolute neutrophil count (ANC) of ≤1.5 x 109 per liter
* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2008-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gino Montagnani, MD, Study Chair — AstraZeneca; Mario diFiorino, Principal Investigator — Ospedale Unico della Versilia (Lido di Camaiore, Lucca Italy)
Locations (21):
- Italy (21):
  - Research Site, Fermo, AP
  - Research Site, Bergamo, BG
  - Research Site, Brindisi, BR
  - Research Site, Carbonia, CA
  - Research Site, Termoli, CB
  - Research Site, Aversa, CE
  - Research Site, Catania, CT
  - Research Site, Nicosia, EN
  - Research Site, Lido di Camaiore, LU
  - Research Site, Messina, ME
  - Research Site, Milazzo, ME
  - Research Site, Monza, MI
  - Research Site, Roma, Roma
  - Research Site, Nocera Inferiore, SA
  - Research Site, Vallo della Lucania, SA
  - Research Site, La Spezia, SP
  - Research Site, Collegno, TO
  - Research Site, Frattaminore
  - Research Site, Lecco
  - Research Site, Palermo
  - Research Site, Partinico

REFERENCES:
- [Derived] Kasper S, Montagnani G, Trespi G, Di Fiorino M. Treatment of depressive symptoms in patients with schizophrenia: a randomized, open-label, parallel-group, flexible-dose subgroup analysis of patients treated with extended-release quetiapine fumarate or risperidone. Int Clin Psychopharmacol. 2015 Jan;30(1):14-22. doi: 10.1097/YIC.0000000000000053. PMID 25356632
- [Derived] Di Fiorino M, Montagnani G, Trespi G, Kasper S. Extended-release quetiapine fumarate (quetiapine XR) versus risperidone in the treatment of depressive symptoms in patients with schizoaffective disorder or schizophrenia: a randomized, open-label, parallel-group, flexible-dose study. Int Clin Psychopharmacol. 2014 May;29(3):166-76. doi: 10.1097/YIC.0000000000000017. PMID 24681810

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult male and female patients. with a diagnosis of schizophrenia or schizoaffective disorder (according to DSM-IVTR criteria). with depressive symptoms HAM-D baseline score ≥ 20. and HAM-D item 1 score ≥2.
Groups:
- Seroquel XR: Seroquel XR dose uptitrated starting from 300 mg in the evening on day 0, then increasing to 600 mg and up to 800 mg in the following two evenings. Previous antipsychotic was taken at the full dose on day 0, half dose on day 1 and stopped from day 2. From day 3 onwards it was possible to adjust the Seroquel XR dose, depending on the clinical response and tolerability of the patient, within the range of 400-800 mg per day
- Risperidone: Risperidone dose was uptitrated starting from 1 mg bid (morning and evening) on day 0, then increasing to 2 mg bid and up to 3 mg in the following two days. As per the other arm, previous antipsychotic was taken at the full dose on day 0, half dose on day 1 and stopped from day 2. From day 2 onwards, it was allowed to adjust he dose of Risperidone depending on the clinical response and tolerability of the patient.
Period: Overall Study
Arm/Group | Seroquel XR | Risperidone
Started | 109 | 107
Completed | 91 | 81
Not Completed | 18 | 26
Not completed — Adverse Event | 8 | 5
Not completed — Lack of Efficacy | 1 | 4
Not completed — Protocol Violation | 2 | 4
Not completed — Withdrawal by Subject | 6 | 10
Not completed — Known risperidone intolerance | 0 | 1
Not completed — Past use of Seroquel -stopped due to AE | 0 | 1
Not completed — Low study drug dose | 0 | 1
Not completed — Glycosylated Hemoglobin >8 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Seroquel XR | Risperidone | Total
Number analyzed (Participants) | 107 | 103 | 210
Age Continuous [Mean (Standard Deviation); unit: years] — Number of participants is lower than number in Participants Flow module. 6 participants, 2 in Seroquel XR and 4 in Risperidone, were not valid for safety population because they did not assume any study drug administration.
  years | 42.46 (10.71) | 42.08 (11.48) | 42.27 (11.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 40 | 91
  Male | 56 | 63 | 119

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 of Calgary Depression Scale for Schizophrenia (CDSS) Score.
Description: The CDSS scale is used to assess the level of depression in schizophrenia and to estimate the severity of depressive symptoms.
  CDSS has 9 items rated on four-point scale: 0=absent; 1=mild; 2=moderate; 3=severe. Anchor point descriptions are provided to aid differentiation between each item score. The first eight items are rated on basis of patients' responses to questions; the 9 item is based on clinician's assessment.
  The sum score is derived by adding the point score of all items (from 0 to 27 points); total score 4-5 is considered for minor depression and 6-7 score for major depression.
Time Frame: 12 week from baseline to last visit
Measure: Least Squares Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Seroquel XR | Risperidone
Number analyzed (Participants) | 107 | 103
Score on a scale | 7.31 (6.1) [6.10 to NA] | 5.53 (6.4) [6.40 to NA]

2. Secondary Outcome: Change From Baseline to Week 12 of HAM-D Score
Description: 21-item scale for depression. Symptoms are rated finely (on a 5-point scale: absent; doubtful or trivial; mild: moderate severe) or coarsely (on a 3- point scale: absent; doubtful or mild; obvious, distinct, or severe).Total score range 0- 66, higher values represent worse outcome.Number of participants refers to valid for efficacy per protocol. Change:total score at week 12 minus total score at baseline.
Time Frame: 12 weeks from baseline to last visit
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Seroquel XR | Risperidone
Number analyzed (Participants) | 107 | 103
Score on scale | -29.83 (10.13) | -23.02 (10.33)

3. Secondary Outcome: Change From Baseline to Week 12 of PANSS Score
Description: 30-item scale where each symptom is rated on a severity ranging from 1-7. Symptoms are categorized into 7 items referring to positive, 7 items referring to negative and 16 general psychotic. Total score range 30- 210, higher values represent worse outcome. Number of participants analyzed refers to valid for efficacy per protocol population.
Time Frame: 12 weeks from baseline to last visit
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Seroquel XR | Risperidone
Number analyzed (Participants) | 107 | 103
score on scale | 102.26 (24.14) | 100.51 (25.65)

4. Secondary Outcome: - Change From Baseline to Week 12 of Clinical Global Impression (CGI- Severity of Illness) Score
Description: The CGI-S subset ranges from 1 to 7 such that a score of 1 indicates "normal, not at all ill", while a score of 7 indicates "among the most extremely ill of patients". The change from start of treatment (baseline V2) in the Severity of Illness will be calculated by subtracting the score at start of treatment (baseline V2) from the following visits
Time Frame: 12 weeks from baseline to last visit
Measure: Least Squares Mean (Standard Deviation); unit: Score on scale
Arm/Group | Seroquel XR | Risperidone
Number analyzed (Participants) | 107 | 103
Score on scale | -1.50 (1.33) [1.33 to NA] | -1.04 (1.31) [1.31 to NA]

5. Secondary Outcome: CGI- Global Improvement Mean Score at Week 12
Description: as for outcome 4
Time Frame: 12week: descriptive statistic of CGI by visit and treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Seroquel XR | Risperidone
Number analyzed (Participants) | 107 | 103
score on a scale | 91 (4.47) [NA to NA] | 88 (4.55) [NA to NA]

6. Secondary Outcome: Change From Baseline to Week 12 of Drug Attitude Inventory 10 Item Scale (DAI 10) Score
Description: These items are presented as self-report statements with which the patient agrees or disagrees. Each response is scored as +1 if correct or -1 if incorrect. The final score is the grand total of the positive and negative points. A positive score means a positive subjective response. A negative total score means a negative subjective response
Time Frame: 12 week from baseline to last visit
Measure: Least Squares Mean (Standard Deviation); unit: score on scale
Arm/Group | Seroquel XR | Risperidone
Number analyzed (Participants) | 107 | 103
score on scale | 86.38 (4.12) [4.12 to NA] | 76.64 (4.70) [4.70 to NA]

7. Secondary Outcome: Change From Baseline in the Simpson Angus Scale (SAS) Total Score to Week 12 as an Indication of Neurological Side Effects Section
Description: Extrapyramidal Side Effects (EPS) will be assessed using the Simpson-Angus Scale (SAS; Simpson GN et al 1970) . The CRF is source data for these assessments and day 0 is considered as baseline.
  The SAS scale, containing 10 items, will be rated on a five-point scale where 0 is normal and 4 are severe symptoms. Min score =0, max score 40
  Change from start of treatment (day 0) will be calculated as the visit score minus the score at start of treatment for each of the neurological assessments.
Time Frame: 12 weeks from baseline to last visit
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Seroquel XR | Risperidone
Number analyzed (Participants) | 107 | 103
score on scale | 2.74 (5.29) | 3.88 (5.24)

8. Secondary Outcome: Concomitant Use of Antidepressive Drugs From Baseline to Week 12
Description: Number of concomitant users of antidepressive drugs during the study; the number of participants analyzed refers to safety population, that is to overall participants excluding 6 participants who did not assume any study drug administration
Time Frame: 12 week from baseline to last visi
Measure: Number; unit: Participants
Arm/Group | Seroquel XR | Risperidone
Number analyzed (Participants) | 107 | 103
Participants | 12 | 11

9. Secondary Outcome: Change From Screening Visit to Week 12 of Prolactin Live
Description: Plasma prolactin live was drawn prior to morning meal at the screening visit at the last visit
Time Frame: 12 week from screening visit to last visit
Measure: Least Squares Mean (Standard Deviation); unit: KG
Arm/Group | Seroquel XR | Risperidone
Number analyzed (Participants) | 107 | 103
KG | 61.20 (29.77) [29.77 to NA] | 90.80 (55.78) [55.78 to NA]

10. Secondary Outcome: Body Mass Index (BMI) at Week 12
Description: Patient weight and height have been be collected in order to assess the Body Mass Index (BMI). The mean BMI values reported are assessed after 12 weeks of treatment.
Time Frame: 12 week
Measure: Mean (Standard Deviation); unit: Kg/m^2
Arm/Group | Seroquel XR | Risperidone
Number analyzed (Participants) | 107 | 103
Kg/m^2 | 29.07 (6.65) | 28.80 (5.31)

11. Secondary Outcome: Concomitant Use of Antidepressive Drugs From Baseline to Week 12
Description: Number of concomitant users of antidepressive drugs during the study; the number of participants analyzed refers to ITT/safety population, that is to overall participants excluding the 6 participants who did not assume any study drug administration
Time Frame: Change of drug use from baseline to last visi
Measure: Number; unit: Participants
Arm/Group | Seroquel XR | Risperidone
Number analyzed (Participants) | 107 | 103
Participants | 14 | 17

ADVERSE EVENTS:
Arm/Group | Seroquel XR | Risperidone
Serious Adverse Events (participants affected / at risk) | 4/109 | 4/107
Other Adverse Events (participants affected / at risk) | 28 | 21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Seroquel XR (N=109) | Risperidone (N=107)
Disorientation (Psychiatric disorders) | 0 | 1
Psycotic Disorder (Psychiatric disorders) | 0 | 1
Delusion (Psychiatric disorders) | 0 | 1
Extrapiramidal Syndrome (Nervous system disorders) | 0 | 1
Faint/Syndrome (Nervous system disorders) | 1 | 0
Acute Psycosis (Psychiatric disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Social Stay Hospitalisation (Social circumstances) | 1 | 0
Cardiocircolatory Arresti (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Seroquel XR | Risperidone
Hyperprolactinemia (Endocrine disorders) | 1/109 | 10/107
Dry Months (Gastrointestinal disorders) | 5/109 | 0/107
Asthenia (General disorders) | 3/109 | 5/107
Weight Increse (Investigations) | 3/109 | 2/107
Sedation (Nervous system disorders) | 5/109 | 1/107
Somnolence (Nervous system disorders) | 6/109 | 2/107
Hypotension (Vascular disorders) | 5/109 | 1/107

LIMITATIONS AND CAVEATS:
Multicentre, randomized, open-label, flexible dose, parallel group, non inferiority

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less